CLINICAL TRIAL: NCT00559117
Title: A Phase I, Open-Label, Dose Ranging Study to Assess the Safety and Distribution of Single or Multiple Doses of VB-111 in Patients With Advanced Metastatic Cancer
Brief Title: A Phase I Study to Assess the Safety and Distribution of VB-111 in Patients With Advanced Metastatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT-111001 (VB-111)
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Advanced and/or Metastatic Solid Organ Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cohort (Experimental)
  Interventions: Drug: VB-111

INTERVENTIONS:
Drug: VB-111 — A single intravenously infusion of diluted VB-111 should be administered 1 ml/minute

SUMMARY:
Aim of the study is to evaluate the safety and find the maximal tolerated dose of VB-111 in Patients with Advanced Metastatic Cancer

DETAILED DESCRIPTION:
Nine Cohorts of dose escalating VB-111 were completed with a total of 56 subjects enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* Histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. For Cohort 8, malignancy will include only NET or RCC.
* Karnofsky performance status of ≥70%
* Patients with an adequate hematological profile
* Patients with an adequate renal function
* Males and Females of childbearing potential must utilize a standard contraception method
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Patients, who suffered from an acute cardiac event within the last 12 months
* Patients with active vascular disease, either myocardial or peripheral
* Patients with proliferative and/or vascular retinopathy
* Patients with known liver disease (alcoholic, drug/toxin induced, genetic, or autoimmune)
* Patients with known CNS metastatic disease
* Patients testing positive to one of the following viruses: HIV, HBV or HCV
* Patients receiving chemotherapy or radiotherapy within the last 4 weeks before enrolment
* Patients that have undergone major surgery within the last 4 weeks before enrolment
* Patients may not have received anti-angiogenic therapy within the previous 8 weeks before enrolment.
* Patients may not have received any other investigational agent within 4 weeks before enrolment.
* Patients with an ongoing requirement for an immunosuppressive treatment, including the use of glucocorticoids or cyclosporin, or with a history of chronic use of any such medication within the last 4 weeks before enrolment
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Triozzi, Dr., Principal Investigator — The Cleveland Clinic; Andrew Brenner, MD, Principal Investigator — UTHSC- CTRC and Institute for Drug Development
Locations (3):
- United States (3):
  - Dana Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - UTHSC- CTRC and Institute for Drug Development, San Antonio, Texas